CLINICAL TRIAL: NCT02998892
Title: Effects of Microbouts of Activity on Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1769
Record Dates: First submitted 2016-12-02; First posted 2016-12-21 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Health Behavior
Keywords: Sedentary Behavior
MeSH Terms: conditions — Health Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Exercise Training (Active Comparator): Participants will be asked to perform moderate-intensity exercise (brisk walking) for 45 minutes for 5 days/week for 6 weeks. This intervention corresponds to the current recommendations.
  Interventions: Behavioral: Traditional Exercise Training
- Daily Microbursts of Activity (Experimental): Participants will be asked to break up their sedentary activities of daily living for 5-minutes every hour for 9 hours, 5 days/week, by brisk walking for 6 weeks.
  Interventions: Behavioral: Daily Microbursts of Activity

INTERVENTIONS:
Behavioral: Traditional Exercise Training — Participants will be asked to perform moderate-intensity exercise (brisk walking) for 45 minutes for 5 days/week for 6 weeks. This intervention corresponds to the current recommendations.
  Arms: Traditional Exercise Training
Behavioral: Daily Microbursts of Activity — Participants will be asked to break up their sedentary activities of daily living for 5-minutes every hour for 9 hours, 5 days/week, by brisk walking for 6 weeks.
  Arms: Daily Microbursts of Activity

SUMMARY:
Population studies suggest that time spent in sedentary behaviors is associated with all-cause mortality including obesity, diabetes, and cardiovascular diseases, independent of time spent in exercise. Frequent interruptions to sedentary time are however beneficially associated with metabolic health outcomes, even in individuals who exercise regularly. The goal is to use integrative approach to understand the biological mechanisms that underlie these associations in a longitudinal intervention study in overweight sedentary adults. The investigators believe that the proposed study will provide an initial evidence base for the health benefits of breaking up prolonged sitting with short bursts of activity. This innovative strategy may be more effective at combating the adverse effects of sedentary behaviors than more traditional approaches.

DETAILED DESCRIPTION:
To compare the effects of 6-weeks of microbursts of moderate-intensity activity to a calorically equivalent single bout of 45 minutes of moderate-intensity exercise training, both performed 5 days per week for a total of 45 minutes, in free-living sedentary overweight adults on:

Aim 1: plasma inflammatory and cardiometabolic health biomarkers in association with total energy expenditure and time spent in sedentary behaviors.

H1: Microbursts of activity will result in higher daily energy expenditure and lower time spent sedentary, as respectively measured with doubly labeled water and accelerometry, than traditional exercise training. This will be associated with healthier inflammatory Interleukin 1 alpha (IL1a), Interleukin 6 (IL6), Interleukin 10 (IL10), Tumour Necrosis Factor alpha (TNFa) and cardiometabolic (triglycerides, cholesterol, C-Reactive Protein (CRP), High-density lipoprotein (HDL), and Low-density lipoprotein (LDL) profiles compared to those obtained with traditional exercise training program.

Aim 2: 24-hr total fat and carbohydrate oxidation, exogenous carbohydrate oxidation, dietary fat trafficking between oxidation and incorporation into muscle lipid fractions, and mitochondrial function.

H2: Both one single continuous bout and microbouts of activity will increase 24-hr total (whole-room calorimetry) and dietary (D31-palmitate) fat oxidation due to greater mitochondrial lipid oxidation (high resolution respirometry) and lower incorporation of dietary fatty acid into muscle lipid fractions (D31-palmitate), as compared to baseline sedentary control condition. Microbouts of activity will further result in greater increases in 24-hr total (whole-room calorimetry) and exogenous (U-13C6 glucose) carbohydrate oxidation and in mitochondrial carbohydrate-linked oxidation, than traditional isocaloric exercise training.

Aim 3: Whole-body insulin sensitivity and daily glucose mean and variability. H3: Both one single continuous bout and microbouts of activity will improve whole-body insulin sensitivity Intravenous Glucose Tolerance Test (IVGTT) compared to the baseline sedentary condition, but the improvement will likely be higher with the microbouts of activity. However, only the microbouts of activity will improve postprandial glycemia and the daily oscillations in glucose level as measured by CGM.

Exploratory aim: Self-perceived appetite and hunger.

ELIGIBILITY:
Inclusion Criteria:

* Overweight but weight stable (+/- 3kg over previous 6 months) sedentary male and female adults (n=30) will be recruited.
* Ages between 18-45 years old
* BMI of 25-35 kg/m2
* Sedentary ( self report < 150min/wk of moderate-to-vigorous activity or less than 6,500 steps per day as measured for 5 days in free-living conditions with a pedometer).
* The use of birth pill control will be accepted

Exclusion criteria:

* Any history of renal (present or past kidney failure, kidney transplant, dialysis or kidney cysts),
* Uncontrolled hypertension
* Cardiovascular (present or past atherosclerosis, heart attack, ischemic stroke, heart failure)
* Hepatic diseases (past or present hepatitis B or C, fibrosis, cirrhosis, NAFLD/NASH)
* Type 1 or 2 diabetes
* Cancer
* Smoking
* Consumption of drugs (marijuana included)
* Consumption of alcohol (>40g/d)
* HIV positivity
* Psychiatric disorders
* Any medications known to interfere with lipid or energy metabolism
* Known physical activity contraindications
* Major illness/physical problems (acute or chronic) that may limit their ability to perform the walking activities

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Changes in sedentary time as measured by ActiPAL | weeks 1-2 and weeks 5-6
  Over each 2 week period, participants will be instructed to wear an ActiPAL (PALTechnologies: Glasgow, Scotland) activity monitor on their right leg. Participants will be instructed to wear the monitors at all times except when sleeping or participating in water-based activities. The time-stamped "event" data file from the activPAL software will be used to determine time spent sitting/lying, standing and stepping per day.
Changes in insulin sensitivity | Week 2 and week 8
  Insulin sensitivity will be determined via an insulin modified frequently sampled intra-venous glucose tolerance test (IVGTT). After baseline samples, intravenous glucose (0.3 g/kg) will be infused over 1 minute, followed by insulin at 0.03 U/kg, 20 minutes after glucose administration. Blood samples will be frequently sampled over 5 hours, and insulin sensitivity will be calculated using the Bergman minimal model.
Postprandial glycemia | Week 2 and week 8
  Incremental area under the curve of plasma glucose concentration measured in fasting and every hour for 14 hours.

SECONDARY OUTCOMES:
Changes in total energy expenditure (TEE) | week 1-2 and week 5-6
  Total energy expenditure (TEE) will be measured before and at the end of the intervention using doubly labeled water (DLW) over a 10-day period, as previously described (31). Subjects will ingest premixed 2g/kg total body water (TBW), estimated as 73% of fat free mass) dose of DLW composed of 0.2 and 0.15 g/kg estimated TBW of H218O and 2H2O, respectively. Urine samples will be collected in duplicate on days 0, 6, 8 and 10. 2H and 18O enrichment will be determined in urine samples by isotope ratio mass spectrometry (Delta V Advantage IRMS)
Changes in Moderate-to-vigorous physical activity as measured by ActiGraph | weeks 1-6
  Over the same 10-day period, participants will be instructed to wear an Actigraph GT3X+ accelerometer (Actigraph, LLC, Fort Walton Beach, FL) on their hip. Participants will be instructed to wear the monitors at all times except when sleeping or participating in water-based activities.
24hr substrate oxidation and energy expenditure | Week 2 and week 8
  Gas exchange are measured for 24hr by whole room calorimetry and nitrogen excretion is measured in the urines collected for 24hr.
  24hr energy expenditure is then calculated using 24hr VCO2, 24hr VO2 and 24hr urinary nitrogen excretion with the Weir equation.
  24hr carbohydrate, fat and protein oxidation are calculated using 24hr VCO2, 24hr VO2 and 24hr urinary nitrogen excretion with the Frayn equation.
Changes in Dietary Carbohydrate Oxidation | week 2 and week 8
  After the investigators have shown the subjects the procedure, subjects will collect their own hourly breath sampling for CO2 by blowing through a straw into two 15ml Vacutainers. Breath CO2 will be sampled directly from the Vacutainer with a syringe, and 13CO2 /12CO2 measured with IRMS.
Changes in Dietary Fat Oxidation | week 2 and week 8
  Hourly urine sampling will be collected by the subjects for 24 hours and stored in 5mL cryovials at -20C until further analysis. To measure 2 hour fat oxidation, 2 hour/1 hour ratios from urine samples will be analyzed, as above described for the doubly labeled water method. The oxidation rate of glucose/water will be calculated from the cumulative recovery of 2 hours in total body water (TBW) as detailed previously.
Postprandial insulinemia | Week 2 and week 8
  Incremental area under the curve of plasma insulin concentration measured in fasting and every hour for 14 hours.
Postprandial NEFA | Week 2 and week 8
  Incremental area under the curve of plasma NEFA as measured in fasting state and every hour for 14 hours.
Postprandial triglyceridemia | Week 2 and week 8
  Incremental area under the curve of plasma TG as measured in fasting state and every hour for 14 hours.
Daily glucose mean and oscillation | Weeks 1-2 and weeks 5-6
  Daily interstitial glucose mean and oscillations as measured by continuous glucose monitoring for 14 consecutive days.
Changes in Mitochondria function | week 2 and week 7
  Freshly isolated skeletal muscle biopsies will be cut into small samples, the fibre bundles separated mechanically and partially teased apart and permeabilised. Small samples (2-5mg) will be added to the 2ml chamber of an Oroboros high-resolution respirometer with a mitochondrial respiration buffer. With the addition of several substrates, different states will be reached to analyse mitochondrial function. Pyruvate, malate and glutamate will be added as substrates to examine respiration through Complex I, succinate will be used to examine respiration through Complex II and octanoylcarnitine will be used to examine respiration through the electron-transferring flavoprotein, ETF.
Changes in plasma inflammatory markers | Week 2 and week 8
  Fasting blood samples will be obtained for the measurements of Interleukin 1 alpha (IL1a), Interleukin 6 (IL6), Interleukin 10 (IL10), Tumour Necrosis Factor alpha (TNFa) and cardiometabolic (triglycerides, cholesterol, C-Reactive Protein (CRP).
changes in plasma total cholesterol, HDL and LDL | Week 2 and week 8
  Fasting plasma blood draw for the measurement of total cholesterol, HDL and LDL.

OTHER OUTCOMES:
Self-perceived appetite and hunger | Week 2 and week 8
  Self-perceived hunger, satiety and prospective food consumption as measured by visual analog scale before and after standard breakfast, lunch, and dinner.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Bergouignan, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No